CLINICAL TRIAL: NCT02358564
Title: Gut Permeability, Sensitivity and Symptomatology: Is There a Link and Explanation for Exacerbation of Symptoms Post Meals
Brief Title: Gut Permeability, Sensitivity and Symptomatology
Acronym: GPSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Erlangen-Nürnberg (Other); Heidelberg University (Other); University of Leeds (Other)
Responsible Party: Principal Investigator, Madhusudan (Madhu) Grover, MBBS, Assistant Professor of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-000837
Record Dates: First submitted 2015-01-30; First posted 2015-02-09 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Irritable Bowel Syndrome; Visceral Hypersensitivity
Keywords: IBS; Irritable Bowel Syndrome; Visceral Hypersensitivity; Permeability; Small Bowel; Lactulose; Mannitol
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (Active Comparator): Participants will receive a Gastrointestinal Permeability Test, Upper Endoscopy, Rectal Barostat and Infusion of Fats.
  Interventions: Procedure: Gastrointestinal Permeability Test; Procedure: Upper Endoscopy; Procedure: Rectal Barostat and Infusion of Fats
- Irritable Bowel Syndrome Patients (Experimental): Participants will receive a Gastrointestinal Permeability Test, Upper Endoscopy, Rectal Barostat and Infusion of Fats.
  Interventions: Procedure: Gastrointestinal Permeability Test; Procedure: Upper Endoscopy; Procedure: Rectal Barostat and Infusion of Fats

INTERVENTIONS:
Procedure: Gastrointestinal Permeability Test — This test will involve ingesting a solution followed by urinalysis
Procedure: Upper Endoscopy
Procedure: Rectal Barostat and Infusion of Fats — Feeding tube will be placed, as well as a small balloon in the rectum.

SUMMARY:
To better understand the relationship between gut barrier function and the symptomatology and pathophysiology of irritable bowel syndrome (IBS).

ELIGIBILITY:
Inclusion criteria

* Age 18 to 70 years
* No abdominal surgery (except appendectomy, cholecystectomy, hernia repair, hysterectomy, and C-section).
* Written informed consent

Exclusion criteria

* Females who are pregnant or breastfeeding
* Use of tobacco products within the past 6 months (since nicotine may affect intestinal permeability)
* Use of NSAIDs or aspirin within the past week (since NSAIDs affect intestinal permeability)
* Use of oral corticosteroids within the previous 6 weeks
* Ingestion of artificial sweeteners such as Splenda (sucralose), Nutrasweet (aspartame), lactulose or mannitol 2 days before the study tests begins, e.g. foods to be avoided are sugarless gyms or mints and diet soda.
* Ingestion of any prescription, over the counter, or herbal medications which can affect gastrointestinal transit 7 days before the study begins.
* Proton pump inhibitors.
* Antibiotics for the preceding 60 days before the start of the study.
* (vii) Alcohol intake beyond the recommended safe limit (<21 unites per week)
* Bleeding disorders or medications that increase risk of bleeding from mucosal biopsies.
* Known allergy to fluorescein
* Inflammatory bowel diseases, celiac disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-02; Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Mean Percent of complete epithelial cell loss | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Madhusudan Grover, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials